CLINICAL TRIAL: NCT01698255
Title: Psychotherapy for Late Life Depression
Acronym: ENGAGE-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1108011880; 11108011880 (Other: WCMC IRB); P30MH085943-05 (NIH)
Record Dates: First submitted 2012-08-02; First posted 2012-10-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Depression
Keywords: Depression; Geriatrics
MeSH Terms: conditions — Depression | interventions — engage 8200

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ENGAGE (Experimental): ENGAGE is a stepped care psychotherapy based on what is known about how older adults respond to depression interventions. Stepped care is a model of treatment that starts with the minimum effective therapeutic techniques first, and then based on how well people respond to treatment, additional therapeutic techniques are added until people are recovered from their depression. The steps of ENGAGE are:
  1. basic social and physical engagement, which has been found to be a very effective depression strategy for most older adults;
  2. the addition of strategies to address clinical features of depression interfering with treatment engagement, namely affect regulation, pessimism, and disorganization.
  Interventions: Behavioral: ENGAGE
- Standard of Care Psychotherapy (Active Comparator): The comparison group for this study will be the current standard of care psychotherapy offered by Westchester Jewish Community Services (WJCS) therapists. This type of psychotherapy is often supportive or eclectic in nature. Therapists will focus on helping the subject to express feelings and focus on strengths and abilities in working through current difficulties and transitions. Therapists assigned to provide standard psychotherapy to eligible participants will receive training and supervision from WJCS staff consistent with agency practice.
  Interventions: Behavioral: Standard of Care Psychotherapy

INTERVENTIONS:
Behavioral: ENGAGE
  Arms: ENGAGE
Behavioral: Standard of Care Psychotherapy
  Arms: Standard of Care Psychotherapy

SUMMARY:
This randomized pilot study will test the feasibility of a behavioral intervention for late life depression. Enrolled participants will receive 9 weeks of a specialized form of psychotherapy we call "ENGAGE" or standard of care psychotherapy. ENGAGE is a stepped care psychotherapy based on what is currently known about older adults' response to depression interventions. Stepped care is a model of treatment that starts with the minimum effective therapeutic techniques first, and then based on how well people respond to treatment, additional therapeutic techniques are added until individuals recover from their depression. The treatment components of ENGAGE were selected to match the most common problems seen in older adults with depression. They include instructing the participant in basic problem solving techniques and encouraging re-engagement in rewarding activities.

Participants will be depressed, older adult clients of Westchester Jewish Community Services or outpatient research subjects recruited by the Cornell Institute of Geriatric Psychiatry. In addition to receiving therapy, study participants will also undergo research assessments at the beginning of the study and then at weeks 6 and 9.

DETAILED DESCRIPTION:
A concern about existing psychotherapies is that, while effective in depression, community clinicians find them difficult to implement in older people, particularly those with medical illnesses or disability. As a consequence evidence-based psychotherapies are utilized by a small number of specialized clinicians and offered to small number of select patients.

ENGAGE approaches these problems with a four prong strategy: 1) It developed a brief treatment program consisting of psychotherapeutic components of known efficacy. 2) Among them, ENGAGE selected components most pertinent to older adults. 3) ENGAGE distilled and simplified these components so that they can be accessible to most depressed older patients and taught to large numbers of clinicians. 4) To further simplify and personalize its administration, ENGAGE relies on a stepped approach focusing on engagement in rewarding social and physical activities (a form of behavioral activation), and when needed, adding techniques for management of emotionality (emotional control), negativity bias, and apathy. The self-correcting and least restrictive nature of stepped care approaches has appeal from patient cost/time efficiency and personalized treatment perspective. This project aims to further develop ENGAGE, to study the feasibility of training professionals (master's level social workers) offering care to depressed elderly patients in the community, to obtain preliminary data of its efficacy compared to community-based therapy (CT), and to prepare for an effectiveness (R01) study.

ELIGIBILITY:
Inclusion Criteria (WJCS Participants):

* Current client of Westchester Jewish Community Services;
* Age 60 years or older;
* Diagnosis of depression as determined by WJCS therapists;
* Command of English sufficient to participate in talking therapy;

Inclusion Criteria (Cornell Participants):

* Age 60 years or older;
* Depression as determined by a Patient Health Questionnaire-9 score of 6 or higher (with at least one item being "depressed mood" or "loss of interest/pleasure");
* Command of English sufficient to participate in talking therapy;

Exclusion Criteria:

* Dementia: Mini Mental State Exam score below 24 or clinical diagnosis of dementia by Diagnostic and Statistical Manual IV;
* High suicide risk, i.e. intent or plan to attempt suicide in near future;
* History of psychiatric diagnoses other than major depressive disorder or generalized anxiety disorder (including bi-polar depression, psychotic depression, schizoaffective disorders).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Depression | 3 months
  To compare the effectiveness of the ENGAGE intervention in reducing depressive symptoms with that of the standard of care psychotherapy. We will assess severity of depression at Baseline. 6 weeks and 3 months using the Hamilton Depression Rating Scale as the primary measure.

CONTACTS AND LOCATIONS:
Overall Officials: George Alexopoulos, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Westchester Jewish Community Services, Hartsdale, New York
  - Weill Cornell Medical College, White Plains, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexopoulos GS, O'Neil R, Banerjee S, Raue PJ, Victoria LW, Bress JN, Pollari C, Arean PA. "Engage" therapy: Prediction of change of late-life major depression. J Affect Disord. 2017 Oct 15;221:192-197. doi: 10.1016/j.jad.2017.06.037. Epub 2017 Jun 19. PMID 28647669
- [Derived] Alexopoulos GS, Raue PJ, Kiosses DN, Seirup JK, Banerjee S, Arean PA. Comparing engage with PST in late-life major depression: a preliminary report. Am J Geriatr Psychiatry. 2015 May;23(5):506-13. doi: 10.1016/j.jagp.2014.06.008. Epub 2014 Jun 26. PMID 25081818